CLINICAL TRIAL: NCT02136342
Title: Phase 1 Trial Evaluating Tolerability and Pharmacokinetics of Chlorogenic Acid for Injection in Patients With Advanced Cancer
Brief Title: Phase 1 Trial of Chlorogenic Acid in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study site change
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Sichuan J.Z. Bio-chemical Science and Technology Development Co., Ltd (Industry)
Responsible Party: Principal Investigator, Shi Yuankai, Dr., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYS-I-01
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Advanced Cancer
Keywords: no available effective treatment
MeSH Terms: interventions — Chlorogenic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chlorogenic acid (Experimental)
  Interventions: Drug: chlorogenic acid

INTERVENTIONS:
Drug: chlorogenic acid

SUMMARY:
The purpose of the study is to explore if chlorogenic acid is safe in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* advanced cancer with no effective treatment
* Karnofsky performance status no less than 70
* adequated organ function
* informed consent

Exclusion Criteria:

* allergic to chlorogenic acid
* persistent toxicities from previous treatment (no less than grade 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-05; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | within the first 60 days after the first dose of chlorogenic acid

SECONDARY OUTCOMES:
dose-limiting toxicity | within the first 30 days after the first dose of chlorogenic acid
maximum tolerated dose | within the first 30 days after the first dose of chlorogenic acid
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of chlorogenic acid | within the first 30 days after the first dose of chlorogenic acid
improvement in cancer-related symptoms and quality of life | within 1 year after the first dose of chlorogenic acid

OTHER OUTCOMES:
Change in number of red blood cell and level of hemoglobin | within 1 year after the first dose of chlorogenic acid
change in the diameters of lymph node metastasis | within 1 year after the first dose of chlorogenic acid
change in levels of tumor markers | within 1 year after the first dose of chlorogenic acid

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Dr., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences